CLINICAL TRIAL: NCT00169390
Title: Comparison of Monoamines Oxidases A and B Activities and the Metabolism of Nicotine in Smoking and Nonsmoking Pregnant Women and in Their Newborns. Evaluation of Their Effects on the Newborns' Behavior
Brief Title: Monoamine Oxidases in Smoking Pregnant Women and Newborns
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Mission Interministérielle de Lutte contre la Drogue et la Toxicomanie (MILDT) (Unknown); Mutuelle Générale de l'Education Nationale (MGEN) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Ivan Berlin, Groupe Hospitalier Pitie-Salpetriere, INSERM U677
Other Study IDs: RBM0344
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2009-08

CONDITIONS: Smoking; Pregnancy; Newborn
Keywords: smoking; pregnancy; newborns; monoamine oxidases
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma DHPG, HVA, 5HIAA, 5HT, cotinine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pregnant smokers
- pregnant non smokers

SUMMARY:
Smoking substantially inhibits the activities of both monamine oxidase (MAO) A and B enzymes.

Aims of this study: to compare MAO activities and nicotine and cotinine in peripheral blood of smoking and nonsmoking pregnant women, in their placenta and in cord blood and relate them with the behavior of their newborns being observed during 48 hours after birth.

DETAILED DESCRIPTION:
40 pregnant smoking and 40 pregnant nonsmoking women will be included at the end of the 2nd trimester.

Assessments: smoking characteristics, plasma cotinine, DHPG, DOPAC, 5HIAA concentrations reflecting MAOA activity and platelet MAOB activity will be measured just after inclusion (end of 2nd trimester), just before delivery in venous maternal blood and just after delivery in cord blood.

The newborns' behavior (wellbeing) will be assessed every 8 hour after birth for 2 days.

Comparisons will be made between smoking and nonsmoking women and their newborns.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy of 5 or 6 months
* nonsmokers: lifetime smoking of less than 100 cigarettes; smokers: unable to stop smoking during the first 3 months of pregnancy; smoking at least 10 cigarettes/day.

Exclusion Criteria:

* pathological pregnancies
* opioid dependence; alcoholism.
* chronic psychiatric, hematological, neurological disorders
* eclampsia
* chronic antidepressant or neuroleptic treatment
* current nicotine replacement therapies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant smoking or not smoking women
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2004-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
monoamine oxidase markers | at birth

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Berlin, MD, PhD, Study Chair — Groupe Hospitalier Universitaire Pitié-Salpêtrière, Service de Pharmacologie and INSERM U677

REFERENCES:
- [Background] Berlin I, Anthenelli RM. Monoamine oxidases and tobacco smoking. Int J Neuropsychopharmacol. 2001 Mar;4(1):33-42. doi: 10.1017/S1461145701002188. PMID 11343627
- [Derived] Berlin I, Heilbronner C, Georgieu S, Meier C, Launay JM, Spreux-Varoquaux O. Reduced monoamine oxidase A activity in pregnant smokers and in their newborns. Biol Psychiatry. 2009 Oct 15;66(8):728-33. doi: 10.1016/j.biopsych.2009.05.029. Epub 2009 Jul 17. PMID 19615672